CLINICAL TRIAL: NCT00580723
Title: Effects of PRK 124 (0.125%) Lotion in Acne Rosacea
Brief Title: Effects of PRK 124 Lotion in Acne Rosacea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: SenetekPLC (Unknown)
Responsible Party: Principal Investigator, Christopher Zachary, MBBS, FRCP, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-5307; Contract SPLC-41239 (Other: University of California, Irvine)
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Acne Rosacea
Keywords: acne; rosacea; acne rosacea; papulopustular rosacea; erythema; telangiectasia; flushing
MeSH Terms: conditions — Rosacea; Acne Vulgaris; Erythema; Telangiectasis; Flushing | interventions — pyratine 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRK 124 (Experimental): Topical PRK 124 (Pyratine-6)(0.125%) moisturizing lotion applied twice daily to the face for 48 weeks. Subjects will wash their faces prior to application. The applications will occur in the mornings and one hour before bedtime.
  Interventions: Other: PRK 124

INTERVENTIONS:
Other: PRK 124 — Topical PRK 124 (0.125%) moisturizing lotion applied twice daily to the face for 48 weeks
  Other Names: Pyratine-6; N-furfuryl-9-(2-tetrahydropyranyl)adenine

SUMMARY:
The purpose of this open-label study is to determine the tolerance and efficacy of twice-daily application of PRK 124 (Pyratine-6)(0.125%) moisturizing lotion for improving the signs and symptoms of mild to moderate facial rosacea.

DETAILED DESCRIPTION:
Cytokinins are plant growth factors that regulate plant growth and differentiation. PRK 124 (N-furfuryl-9-(2-tetrahydropyranyl) adenine)(Pyratine 6™) is a cytokinin that has been shown to have modulatory, anti-ROS (reactive oxygen species), and antisenescence effects on the growth of human skin cells.

Recent clinical studies showed that PRK 124 (0.1%) treatment in 40 subjects for 12 weeks improved the appearance of photodamaged facial skin by decreasing fine wrinkles, roughness and mottled hyperpigmentation. Treatment with PRK 124 lotion furthermore decreased skin transepidermal water loss and also increased skin moisture content. The topical PRK 124 lotion was well tolerated by the subjects with no significant increase in erythema or irritation. Treatment with PRK 124 was shown to decrease both acne and erythema observed at baseline.

Rosacea is a common, chronic dermatosis that is characterized by papules and pustules, persistent erythema and telangiectasia. The objective of this study is to compare the long-term efficacy and tolerance of PRK 124 (0.125%) moisturizing lotion applied twice daily for 48 weeks for improving the clinical signs and symptoms of inflammatory acne rosacea as well as cutaneous signs of skin photodamage.

Study Design:

Twenty four volunteers with mild-to-moderate facial rosacea will participate in this single center, open-label study designed to evaluate the subject=s tolerance and effectiveness of PRK 124 (0.125%) moisturizing lotion applied twice daily for 48 weeks, for improving the signs and symptoms of acne rosacea. Subjects will apply the test lotion twice daily, once in morning and again in the evening before bedtime. Subjects will be assessed at baseline and at 4, 8 and 12 weeks after treatment for improvement in the clinical signs and symptoms of acne rosacea and effect of treatments on transepidermal water loss (TEWL). In addition, the subject's tolerance will be assessed at each follow-up visit (weeks 4, 8, and 12). Facial photographs will be obtained at baseline and at 4, 8 and 12 weeks. Subjects will then be given the opportunity to continue treatment for 36 additional weeks. Subjects must have normal clinical laboratory tests, and if female, a negative urine pregnancy test at 12 weeks to continue the 36 weeks treatment. Clinical laboratory tests and urine pregnancy test will be repeated at week 48 or early study completion. Clinical assessments will be done at weeks 24, 36 and 48 during the last 36 weeks. Additional objective measures of skin moisture content and skin erythema using a chromameter will be done at week 12 and at follow-up visits (weeks 24, 36 and 48). Telephone follow-up will be done at weeks 16, 20, 28, 32 and 40 to assess subject tolerance and compliance.

Primary Study Variables:

The primary study variables are:

Observations by Investigator:

* Inflammatory lesion count
* Erythema and telangiectasia severity
* Global assessment of severity
* Overall improvement over baseline
* Photodamage (fine wrinkles, texture, mottled hyperpigmentation)
* Transepidermal water loss (TEWL)
* Skin moisture content
* Skin erythema as measured by a chromameter

Subject self assessment:

* Signs & symptoms (burning/stinging, erythema/telangiectasia, papules/pustules)
* Overall improvement over baseline
* Photodamage (fine wrinkles, texture, mottled hyperpigmentation)
* Cosmetic acceptability

The local skin tolerance of the treatments will be assessed by the Investigator and by the subject.

ELIGIBILITY:
Inclusion Criteria:

* be at least 21 years old
* be in reasonably good health as defined by the study doctor
* have routine laboratory tests to evaluate your blood cell count, and kidney and liver function
* for females of child-bearing age, not be pregnant or nursing and have a negative urine pregnancy test (except if surgically sterile or at least 1 year menopausal)
* for females, agree to use medically acceptable forms of birth control throughout the entire study (medically acceptable forms of birth control include oral contraceptive ["the pill"], implants such as Norplant®, injectable progesterone [Depo-provera®], diaphragm and spermicide or condoms and spermicide)
* must have mild to moderate acne rosacea
* be willing to refrain from using non-approved lotions, moisturizer, cleansers or lotions on affected facial areas during the treatment period
* be capable of understanding and giving written, voluntary informed consent before study screening
* be willing to consent to facial photographs at baseline and each follow-up visit to monitor treatment with the test product.

Exclusion Criteria:

* have a history or evidence of any chronic or reoccurring skin disease or disorder (e.g., psoriasis, eczema, etc.) affecting the face
* have known or suspected hypersensitivity to study treatment or any of its ingredients
* have used systemic retinoids within 6 months prior to study entry (e.g., acitretin, isotretinoin)
* have received treatment with systemic corticosteroids (e.g. prednisone) or antibiotics within 1 month
* have used topical treatment to the face with retinoids (e.g. tretinoin, adapalene), or antibiotics or corticosteroids, within 2 weeks prior to study entry
* are unwilling to use a sunscreen with an SPF of 30 during the study
* have participated in any clinical trial involving an investigational drug or cosmetic product or procedure within the past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald D Weinstein, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Dermatology Clinical Research Center, Irvine, California, United States

REFERENCES:
- [Background] Verbeke P, Siboska GE, Clark BF, Rattan SI. Kinetin inhibits protein oxidation and glycoxidation in vitro. Biochem Biophys Res Commun. 2000 Oct 5;276(3):1265-70. doi: 10.1006/bbrc.2000.3616. PMID 11027621
- [Background] Wu JJ, Weinstein GD, Kricorian GJ, Kormeili T, McCullough JL. Topical kinetin 0.1% lotion for improving the signs and symptoms of rosacea. Clin Exp Dermatol. 2007 Nov;32(6):693-5. doi: 10.1111/j.1365-2230.2007.02513.x. Epub 2007 Sep 14. PMID 17868391
- See also: UC Irvine Department of Dermatology — http://www.dermatology.uci.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical PRK 124: Topical PRK 124 (Pyratine-6)(0.125%)
Period: Overall Study
Arm/Group | Topical PRK 124
Started | 24
Completed | 16
Not Completed | 8
Not completed — Did not want to participate in extension | 3
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Topical PRK 124
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Erythema Severity
Description: Measured by percent improvement on a scale of 0-4. Subjects received a 0 for no improvement, 1 for less than twenty-five percent improvement, a 2 for twenty-five to fifty percent improvement, a 3 for fifty to seventy-five percent improvement and a 4 for greater than seventy-five percent improvement. Mean scores from all continuing 16 participants were averaged for each encounter, for a total of 8 visits. The percent improvement in mean erythema severity was calculated by comparing the change in mean scores at week 48 to mean scores assessed at baseline.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Population: We had a total of 24 subjects. Five were lost to follow up and three did not want to participate in the extension period. The results from the remaining 16 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: Erythema percent improvement
Arm/Group | Topical PRK 124
Number analyzed (Participants) | 16
Erythema percent improvement | 44.53 (0.68)

2. Secondary Outcome: Skin Tolerance
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Reporting Status: Not Posted

3. Secondary Outcome: Skin Photodamage
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Reporting Status: Not Posted

4. Secondary Outcome: Transepidermal Water Loss (TEWL)
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Reporting Status: Not Posted

5. Secondary Outcome: Cosmetic Acceptability
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Reporting Status: Not Posted

6. Primary Outcome: Inflammatory Lesion Count
Description: Lesion counts were numerically summed for each patient at each encounter, and the average lesion count was calculated from all continuing 16 subjects at each visit, for a total of 8 visits. Percent improvement (reduction in lesion number) was assessed by comparing the average number of lesions at week 48 to the average number of lesions assessed at baseline.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change in number of lesions
Arm/Group | Topical PRK 124
Number analyzed (Participants) | 16
Percent change in number of lesions | 89 (0.58)

7. Primary Outcome: Telangiectasia Severity
Description: Measured by percent improvement on a scale of 0-4. Subjects received a 0 for no improvement, 1 for less than twenty-five percent improvement, a 2 for twenty-five to fifty percent improvement, a 3 for fifty to seventy-five percent improvement and a 4 for greater than seventy-five percent improvement. Mean scores from all continuing 16 participants were averaged for each encounter, for a total of 8 visits. The percent improvement in mean telangiectasia severity was calculated by comparing the change in mean scores at week 48 to mean scores assessed at baseline.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 24, 36, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Telangiectasia percent improvement
Arm/Group | Topical PRK 124
Number analyzed (Participants) | 16
Telangiectasia percent improvement | 27.88 (0.62)

ADVERSE EVENTS:
Arm/Group | Topical PRK 124
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No